CLINICAL TRIAL: NCT03609866
Title: the Effects of Manual Thoracic Compression Technique in Intracranial Pressure in Mechanically Ventilated Patients With Acute Cerebral Injury
Brief Title: Chest Physiotherapy Effects on Intracranial Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Santiago de Compostela (Other)
Responsible Party: Principal Investigator, ricardo miguel rodrigues gomes, principal investigator, University of Santiago de Compostela
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: Usantiago Doct
Record Dates: First submitted 2018-07-10; First posted 2018-08-01 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Acute Brain Injury
Keywords: intracranial pressure increase; chest physiotherapy; ventilated patients; mechanical ventilation
MeSH Terms: conditions — Brain Injuries; Intracranial Hypertension

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Active Comparator): will be performed inferior limbs passive mobilization
  Interventions: Procedure: inferior limb passive mobilization
- experimental (Experimental): rapid thoracic compression technique will be applied
  Interventions: Procedure: rapid thoracic compression technique

INTERVENTIONS:
Procedure: rapid thoracic compression technique — in the expiratory time of the ventilation set, it will be applied a rapid thoracic compression
  Arms: experimental
Procedure: inferior limb passive mobilization — it will be performed a passive mobilization technique on the patient
  Arms: control

SUMMARY:
The investigators will study the effects of a chest physiotherapy technique (rapid thoracic compression) on the intracranial pressure of individuals with acute cerebral injury and with need of intubated mechanical ventilation

DETAILED DESCRIPTION:
Patients with acute brain injury often require invasive mechanical ventilation connection, increasing the risk of developing complications such as respiratory secretions retention. Thethoracic compression is a manual chest physiotherapy technique that can improve clearance of secretions in these patients. Although today the scientific evidence is contradictory, the manual abdomino-thoracic compression may be associated with increased intracranial pressure in patients with acute brain injury.

Objectives: The aim of this work to study the effects of manual thoracic compression technique in intracranial pressure in mechanically ventilated patients. Furthermore, the effects of the technique in different volumes and flows recorded by the ventilator and the relationship between the pressure applied in the intervention group and the different variables will also be studied.

Methodology: It will be a randomized clinical trial, single-blind in the application of the techniques. Patients with acute brain injury in invasive mechanical ventilation will be included, randomized into two groups. In the control group, a technique of passive inferior limbs mobilization will be applied and in the intervention group it will be performed the manual thoracic compression technique. The data of the primary variable, intracranial pressure will be collected with a monitoring system and continuous recording (Integra Camino).

A descriptive analysis of the values collected from the variables in the study will be performed, studying the measures of central tendency. In the presence of normal distribution will be presented mean and standard deviation, and median and interquartile range in case of non-observation of normal distribution. The normality of the samples will be verified with the Kolmogorov-Smirnov test. The verification of the hypothesis in study will be assessed using the Student T test for independent samples in case of sample normality and by the Wilcoxon test otherwise. A multiple linear regression analysis will be performed: considering as a dependent variable the differences in intracranial pressure, difference or volume / minute gain and expiratory flow and between the covariates, the type of technique, the pressure applied in the technique under study, the type of brain injury, age, sex, etc.

ELIGIBILITY:
Inclusion Criteria:

* intubated patients for 48 hours in vc, pc, vcrp
* hemodynamically stable (MAP>60mmHg)
* respiratory stability (PEEP<15cmH2O and FiO2<60%)
* ICP stable (0<icp<20mmHg)
* RASS of 5
* informed consent signed

Exclusion Criteria:

* thoracic fractures
* abdominal injuries that limits local pressure
* systemic or local changes that undergoes with abdominal volume increase
* inferior limbs fractures that contraindicates passive mobilization techniques

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
intracranial pressure changes | 5 minutes before start procedure, immediately after procedure, 5 minutes after the end of procedure and 10 minutes after the end of procedure
  with Camino ICP monitoring

SECONDARY OUTCOMES:
oxygen saturation changes | 5 minutes before start procedure, immediately after procedure, 5 minutes after the end of procedure and 10 minutes after the end of procedure
  with philips monitoring device
peak expiratory flow changes | all the respiratory cycles will be recorded 30 seconds before procedure and during the procedure
  with maquet servo u and servo i ventilators, the purpose is to identify the best peak expiratory flow before and during the procedure, and to compare them.
heart rate changes | 5 minutes before start procedure, immediately after procedure, 5 minutes after the end of procedure and 10 minutes after the end of procedure
  with philips monitoring device
cerebral perfusion pressure changes | 5 minutes before start procedure, immediately after procedure, 5 minutes after the end of procedure and 10 minutes after the end of procedure
  with philips monitoring device

CONTACTS AND LOCATIONS:
Overall Officials: ricardo m rodrigues gomes, PT MSc, Principal Investigator — University of Santiago de Compostela
Locations (1):
- Hospital Álvaro Cunqueiro, Vigo, Galicia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rodrigues-Gomes RM, Prieto Campo A, Martinez Rolan R, Gelabert-Gonzalez M. Effects of rapid chest compression technique on intracranial and cerebral perfusion pressures in acute neurocritical patients: a randomized controlled trial. Crit Care. 2025 Apr 23;29(1):159. doi: 10.1186/s13054-025-05405-8. PMID 40270039
- [Derived] Rodrigues-Gomes RM, Marti JD, Rolan RM, Gelabert-Gonzalez M. Rapid chest compression effects on intracranial pressure in patients with acute cerebral injury. Trials. 2022 Apr 15;23(1):312. doi: 10.1186/s13063-022-06189-w. PMID 35428364